CLINICAL TRIAL: NCT02596659
Title: Effectiveness of Radial Extracorporeal Shockwave Therapy on Tennis Elbow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RESWTonLE201309
Record Dates: First submitted 2015-10-22; First posted 2015-11-04 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-10

CONDITIONS: Lateral Epicondylosis; Lateral Epicondylitis; Tennis Elbow
Keywords: lateral epicondylosis; lateral epicondylitis; shockwave; sonoelastography; tennis elbow; pain intensity; grip strength; upper limb function; stiffness of common extensor tendon
MeSH Terms: conditions — Tennis Elbow; Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The experimental group (Experimental): Participants in the experimental group received radial extracorporeal shock wave therapy (rESWT) plus physical therapy for 3 weeks.
  Interventions: Procedure: Radial extracorporeal shock wave therapy (rESWT); Procedure: Physical therapy
- The control group (Sham Comparator): Participants in the control group received sham shockwave therapy plus physical therapy for 3 weeks.
  Interventions: Procedure: sham shockwave therapy; Procedure: Physical therapy

INTERVENTIONS:
Procedure: Radial extracorporeal shock wave therapy (rESWT) — Each participant in the experimental group received rESWT for 3 sessions, consisting of 2000 impulses for each session, and one session per week over 3 weeks (a total of 6000 shock waves were given). The pneumatic pressure was set at the maximum level tolerable for each patient. The frequency of pulses was set at 10 Hz.
  Arms: The experimental group
Procedure: sham shockwave therapy — Sham shockwave therapy were given by the same physiatrist using the same machine as the experimental group, with the same rESWT protocol (3 sessions, 2000 impulses for each session, one session per week over 3 weeks) and the same frequency (10 Hz) of impulses, but the pneumatic pressure was set at 0.1 bar, with a similar sound to the regular rESWT but without actual energy conduction.
  Arms: The control group
Procedure: Physical therapy — The physical therapy program was performed 3 times a week over the same 3 weeks as rESWT, and consisted of 5 minutes of ultrasound diathermy, 15 minutes of transcutaneous electrical nerve stimulation (TENS), and 10 minutes of therapeutic exercise, including wrist common extensor stretching and self-massage.

SUMMARY:
Background:

Tennis elbow, also known as lateral epicondylitis, is the inflammatory status of insertion site of common extensor tendon to humerus. It is usually related to overuse of local muscle. Radial extracorporeal shock wave therapy (rESWT) is a non-invasive physical treatment. It applies shockwave energy to the lesion site, enhancing the growth of microvascularity, inducing tissue repair, and thus relieving the symptom.

The purpose of this study is to understand the therapeutic effect of rESWT to tennis elbow.

Material and Methods

* Subjects: 30 patients will be recruited from outpatient department of physical medicine and rehabilitation department.
* Duration: 2013.09.01-2015.05.31
* Methods: The patients will be randomly divided into the experimental group and the control group through the draw, with 15 patients in each group. Patients in the experimental group receive rESWT plus routine rehabilitation program. Patients in the control group receive sham shockwave therapy plus routine rehabilitation program.
* Assessment: Before the therapy starts, patients who match the inclusion criteria will be evaluated using tools mentioned below:
* General data: age, sex, body height, body weight, affected side, medical history
* Assess upper extremity function and symptom with Disabilities of the Arm, Shoulder and Hand Questionnaire (DASH)
* Assess severity of pain with Visual Analogue Scale (VAS)
* Assess grip strength with grip strength dynamometer
* Measure the size of tear (if any) of common extensor tendon through ultrasonography, and assess the texture of common extensor tendon through real-time sonoelastography (RTS)

Patients will be followed up 6 weeks, 3months, and 6 months after therapy starts. They will be re-assessed of upper extremity function and symptom, severity of pain, grip strength, and presentation on ultrasonography and RTS.

ELIGIBILITY:
Inclusion Criteria:

* Aged > 18 years old
* Lateral elbow pain lasting > 3 months
* Pain induced by direct compression on the lateral epicondyle or common extensor tendon, resistant wrist extension and pronation in the elbow extension position, or static stretching of common extensor tendon through the palmer flexion in wrist pronation and elbow extension position

Exclusion Criteria:

* Generalized inflammatory arthritis (e.g., rheumatic arthritis)
* Pain at the proximal part of involved arm (e.g., shoulder pain, neck pain)
* Pain other than elbow pain at the involved arm
* Abnormal neurogenic symptom over the involved arm (e.g., radicular pain, hands numbness, hemiplegia)
* Wound or skin lesion at the elbow of the involved arm
* Pregnancy
* Severe local or systemic infection
* Malignancy
* Coagulopathy
* Cardiac pacemaker
* History of surgical treatment at the elbow of the involved arm
* Non-steroid anti-inflammatory drug (NSAID) use orally or topically at the elbow of the involved arm in the past week
* Local steroid injection at the elbow of the involved arm in the past 3 months
* Oral steroid use in the past 6 weeks
* Refusal to sign the informed consent
* Impairment in self-expression (e.g., dementia, aphasia)
* Inability/unwillingness to participate in all the measurements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Changes in pain intensity | At baseline, 6 weeks, 12 weeks and 24 weeks
  Participants were asked to rate their present pain intensity, as caused by the tennis elbow, from 0-10 using the Visual Analogue Scale (VAS). If participants had bilateral tennis elbow, the side with the worse pain intensity was chosen for the assessment.
Changes in grip strength | At baseline, 6 weeks, 12 weeks and 24 weeks
  Maximal grip strength of the involved arm was assessed using a grip strength dynamometer. Participants were asked to grip the dynamometer 3 times, at 15- second rest intervals, and the highest grip strength number was recorded.
Changes in upper limb function | At baseline, 6 weeks, 12 weeks and 24 weeks
  Upper extremity disability and symptoms were assessed using the Taiwan version Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire.
Changes in stiffness of common extensor tendon | At baseline, 6 weeks, 12 weeks and 24 weeks
  The changes in stiffness of common extensor tendon were assessed with sonoelastography. The images of sonoelastography were interpreted with the modified RTS scoring system and analyzed with color histogram.

SECONDARY OUTCOMES:
Changes in size of tear within common extensor tendon | At baseline, 6 weeks, 12 weeks and 24 weeks
  On the 2-D image, the common extensor tendon was located. If there was tear within common extensor tendon, diameters in the 3-D dimension were measured and the size of the tear was calculated as a spheroid.

CONTACTS AND LOCATIONS:
Overall Officials: Tsung-Hsun Yang, MD, Principal Investigator — Kaohsiung Chang Cung Memorial Hospital
Locations (1):
- Department of Physical Medicine and Rehabilitation, Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Khoury V, Cardinal E. "Tenomalacia": a new sonographic sign of tendinopathy? Eur Radiol. 2009 Jan;19(1):144-6. doi: 10.1007/s00330-008-1112-9. Epub 2008 Aug 2. PMID 18677489
- [Background] De Zordo T, Lill SR, Fink C, Feuchtner GM, Jaschke W, Bellmann-Weiler R, Klauser AS. Real-time sonoelastography of lateral epicondylitis: comparison of findings between patients and healthy volunteers. AJR Am J Roentgenol. 2009 Jul;193(1):180-5. doi: 10.2214/AJR.08.2020. PMID 19542412
- [Background] Kwon DR, Park GY, Lee SU, Chung I. Spastic cerebral palsy in children: dynamic sonoelastographic findings of medial gastrocnemius. Radiology. 2012 Jun;263(3):794-801. doi: 10.1148/radiol.12102478. Epub 2012 Apr 10. PMID 22495685
- [Background] Ahn KS, Kang CH, Hong SJ, Jeong WK. Ultrasound elastography of lateral epicondylosis: clinical feasibility of quantitative elastographic measurements. AJR Am J Roentgenol. 2014 May;202(5):1094-9. doi: 10.2214/AJR.13.11003. PMID 24758665
- [Background] Speed C. A systematic review of shockwave therapies in soft tissue conditions: focusing on the evidence. Br J Sports Med. 2014 Nov;48(21):1538-42. doi: 10.1136/bjsports-2012-091961. Epub 2013 Aug 5. PMID 23918444
- [Background] Spacca G, Necozione S, Cacchio A. Radial shock wave therapy for lateral epicondylitis: a prospective randomised controlled single-blind study. Eura Medicophys. 2005 Mar;41(1):17-25. PMID 16175767
- [Background] Ilieva EM, Minchev RM, Petrova NS. Radial shock wave therapy in patients with lateral epicondylitis. Folia Med (Plovdiv). 2012 Jul-Sep;54(3):35-41. doi: 10.2478/v10153-011-0095-5. PMID 23270205
- [Background] Gunduz R, Malas FU, Borman P, Kocaoglu S, Ozcakar L. Physical therapy, corticosteroid injection, and extracorporeal shock wave treatment in lateral epicondylitis. Clinical and ultrasonographical comparison. Clin Rheumatol. 2012 May;31(5):807-12. doi: 10.1007/s10067-012-1939-y. Epub 2012 Jan 27. PMID 22278162